CLINICAL TRIAL: NCT02732795
Title: Effects of Obstructive Sleep Apnea Syndrome and Obesity on Morphine Pharmacokinetics in Children
Brief Title: Sleep Apnea and Obesity Affects on Morphine Pharmacokinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00034512
Record Dates: First submitted 2016-02-04; First posted 2016-04-11 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Pediatric Sleep Apnea; Obesity; Morphine Metabolism
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Morphine dosing (Experimental): Evaluating morphine pharmacokinetics (PK) in 3 groups: normal controls, children with severe OSAS, and obese children with OSAS. Morphine is dosed on ideal body weight in obese children, as recommended by manufacturer. Biomarkers were taken from patients to evaluate their relation to changes in morphine PK.
  Interventions: Other: Morphine pharmacokinetic evaluation

INTERVENTIONS:
Other: Morphine pharmacokinetic evaluation — Each group received morphine and blood drawn to evaluate morphine PK

SUMMARY:
Adenotonsillectomy (AT) is one of the most common pediatric surgeries performed, and is estimated to comprise 530,000 procedures in children under 15 years of age. Historically, the leading cause for these procedures was recurrent infections; however, more recently surgical indications include sleep disordered breathing and obstructive sleep apnea (OSAS). Pre-operative polysomnography (PSG) is recommended for all children with suspected OSAS prior to undergoing AT, although it is unclear whether sleep disordered breathing characteristics predict post-operative outcomes or complications.

Obesity has become an epidemic in the pediatric population. More recently, an increased population of obese children are presenting for AT with upper airway obstruction with or without tonsillar hypertrophy, which is similar to the adult etiology of OSAS. Obesity is a multisystem disease, causing fatty liver and cardiac disease, defects in glucose metabolism, insulin resistance, leptin resistance, and creates a state of chronic inflammation. Markers for inflammation, including tumor necrosis factor (TNF)-α, C-reactive protein (CRP), leptin, interleukin (IL)-6 and IL-10, are abnormal in obese patients and have also been linked to more severe OSAS disease in children even after controlling for BMI.

In pediatrics, medication dosing is based on an actual body-weight calculation, however, recent reports suggest that this dosing method is over-dosing patients with obesity. Therefore, increased respiratory complications after surgery may be related to inappropriate intra-operative opioid dosing.

Specific Aim 1 (SA1): To compare morphine pharmacokinetics in normal children <=12 years of age, non-obese children with severe OSAS, and obese children with severe OSAS. The investigators hypothesize that obesity independently enhances morphine pharmacokinetics.

Specific Aim 2 (SA2): To determine whether biomarkers related to obesity, chronic inflammation, and OSAS predict changes to morphine pharmacokinetics. The investigators hypothesize that inflammatory and obesity-related biomarkers are elevated in overweight children with OSAS, more so in obese children with OSA, compared to lean children with OSAS. In addition, the investigators hypothesizes that leptin independently is linked to altered morphine pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Child presenting for surgery that will require opioids
* Age between 5 -12 years of age

OSAS group:

* Pre-operative polysomnography study conducted prior to day of surgery

Obese:

* Body weight >95th percentile for age.

Exclusion Criteria:

* Emergency procedures involving AT, including tonsillar bleeding
* Patients allergic to morphine
* Patients with comorbidities altering opioid metabolism (i.e. liver disease)
* Patients with chronic inflammatory, rheumatologic, or other confounding co-morbid diseases (i.e. Crohns disease, ulcerative colitis, sickle cell, Sjogren's, etc.)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Plasma Morphine Area Under the Curve (AUC) | Through study completion, up to 24 hours after study initiation
  To determine changes in morphine AUC due to obesity and OSAS
Maximum Plasma Morphine Concentration (Cmax) | Through study completion, up to 24 hours after study initiation
  To determine changes in morphine Cmax due to obesity and OSAS
Time to Maximum Plasma Morphine Concentration (Tmax) | Through study completion, up to 24 hours after study initiation
  To determine changes in morphine Tmax due to obesity and OSAS
Half Life of Plasma Morphine Concentration (T1/2) | Through study completion, up to 24 hours after study initiation
  To determine changes in morphine T1/2 due to obesity and OSAS
Plasma Morphine Clearance (Cl) | Through study completion, up to 24 hours after study initiation
  To determine changes in morphine Cl due to obesity and OSAS
Plasma Morphine Volume of Distribution (Vd) | Through study completion, up to 24 hours after study initiation
  To determine changes in morphine Vd due to obesity and OSAS
Plasma Morphine 3-glucuronide (M3G) Maximum Plasma Concentration (Cmax) | Through study completion, up to 24 hours after study initiation
  To determine changes in M3G Cmax due to obesity and OSAS
Time to Maximum Morphine 3-glucuronide (M3G) Concentration (Tmax) | Through study completion, up to 24 hours after study initiation
  To determine changes in M3G Tmax due to obesity and OSAS
Morphine 3-glucuronide (M3G) to Morphine ratio | Through study completion, up to 24 hours after study initiation
  To determine changes in metabolism of morphine due to obesity and OSAS
Morphine 3-glucuronide (M3G) to Morphine 6-glucuronide (M6G) ratio | Through study completion, up to 24 hours after study initiation
  To determine changes in metabolism of morphine due to obesity and OSAS

SECONDARY OUTCOMES:
Biomarker concentrations | Through study completion, up to 24 hours after study initiation
  To determine whether inflammatory biomarkers correlate to the severity of sleep apnea. Biomarkers that will be studied include IL 1,6,10, CRP, TNF-alpha, leptin, and insulin.

CONTACTS AND LOCATIONS:
Locations (1):
- Bloomberg Children's Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No